CLINICAL TRIAL: NCT05155527
Title: A Phase 2 Double-blind Randomized Placebo-controlled Trial to Assess the Efficacy of Ivermectin in Combination With Favipiravir in Mild-to-moderate COVID-19 Adult Patients
Brief Title: Ivermectin With Favipiravir in Mild-to-moderate COVID-19 Patients
Acronym: IFCOV
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: Prince of Songkla University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CREC067/64BR-MED46
Record Dates: First submitted 2021-12-09; First posted 2021-12-13 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
Keywords: COVID-19; Favipiravir; Ivermectin
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Favipiravir plus Ivermectin (Experimental): Ivermectin 600 mcg/kg once daily for 5 days in combination with Favipiravir for 5-10 days (1,800 mg twice a day in day 1 then 800 mg twice a day for the other days. For BW > 90 kg: 2,400 mg twice a day in day 1 then 1,000 mg twice a day for the other days).
  Interventions: Drug: Ivermectin Tablets
- Favipiravir plus Placebo (Placebo Comparator): Matching placebo once daily for 5 days in combination with Favipiravir for 5-10 days (1,800 mg twice a day in day 1 then 800 mg twice a day for the other days. For BW > 90 kg: 2,400 mg twice a day in day 1 then 1,000 mg twice a day for the other days).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ivermectin Tablets — 6 mg/tablet
  Arms: Favipiravir plus Ivermectin
Other: Placebo — The placebo has same form as Ivermectin.
  Arms: Favipiravir plus Placebo

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infections are rapidly spreading worldwide and continue to be a global public health crisis. The use of repurposed drugs with the potential to inhibit SARS-CoV-2 could be a vital alternative approach when the novel therapeutic has not yet available. The guidelines for emergency treatment of COVID-19 vary across different countries and largely rely on the off-label prescription of repurposed drugs. As a result, clinical studies to generate robust efficacy data for these repurposed drugs are warranted to effectively fight against the ongoing COVID-19 pandemic.

The broad spectrum antiparasitic drug ivermectin has previously been shown to exhibit broad antiviral activities against many RNA and DNA viruses. It has a reliable safety profile with comprehensive data for decades especially in mass drug administration programs for river blindness prophylaxis in several countries in Africa. Owing to its strong inhibitory activity against the replication of SARS-CoV-2 in vitro and its putative role in reducing cytokine storm, the drug has been repurposed to treat COVID-19 patients and has shown promising results in several clinical studies. Ivermectin has thus gained a considerable attention as a potential treatment for COVID-19. However, the National Institute of Health (NIH) and World Health Organization (WHO) currently state that studies on using ivermectin to treat COVID-19 patients remain inconclusive due to insufficient data. Therefore, a large well designed randomized, double blinded, placebo-controlled trial to assess the efficacy of ivermectin is urgently needed.

Another important treatment option for COVID-19 is favipiravir, an antiviral drug for influenza treatment. Although the drug has not been approved for a COVID-19 treatment by the US-FDA, it has been included in Guidelines on clinical practice, diagnosis, treatment, and prevention of healthcare-associated infection for COVID-19 in Thailand. Favipiravir, a known inhibitor of RNA-dependent RNA polymerase, was shown to have an in vitro activity against SARS-CoV-2. The meta-analysis showed a significant improvement in clinical outcome at day 14 along with chest imaging in the favipiravir group compared to standard care. However, there are no significant differences in terms of clinical deterioration rates, viral clearance, oxygen support requirement and side effect profiles. There are still ongoing clinical trials assessing the effectiveness of favipiravir in the treatment of COVID-19.

Antivirals can be generally divided into direct-acting antivirals (DAA) and host-targeting drugs. For example, the widely used drug remdesivir repurposed to treat COVID-19 is a DAA, and chloroquine is considered a host-targeting drug. Because these repurposed drugs were not specifically designed and developed for COVID-19, they are likely to be less efficacious, and partner drugs need to be further explored. Finding a right combination for DAA is a common practice for developing virus treatment regimens. Relying on different modes of action and absence of unfavorable drug interaction, the combinations are usually additive or synergistic. It is important to note that our in vitro data demonstrated the synergistic profile for the combination of favipiravir and ivermectin against SARS-CoV-2. It resulted in 4-fold reduction in the half maximal inhibitory concentration (IC50) as compared to individual drugs, from 1.2 µM to 0.3 µM with a peak Loewe synergy score of over 33.2 and a mean score of 18.8 (noted that Loewe synergy score > 10 indicates synergistic effect).

In response to this COVID-19 pandemic crisis, especially in a resource limited setting like Thailand, clinical studies to evaluate affordable and implementable interventions are a priority and are urgently needed. Ivermectin, a cheap and safe drug, has been widely used in humans for decades, and it has also demonstrated an inhibitory effect against SARS-CoV-2 in vitro. Here, we aim to conduct a multi-center, double-blind, randomized controlled trial in Thailand to reveal the effectiveness of ivermectin as a combination therapy with favipiravir (standard treatment) for COVID-19. The results of this study will provide much needed information for pursuing larger efficacy clinical trials to confirm whether the combination could be effectively used to treat COVID-19. Also, they could provide information on the rate of viral clearance, the primary endpoint of this study, which was proposed to be a predictive surrogate of clinical benefits and used as a proper endpoint in the phase II trials for candidate drug screening for COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient age between 18-65 years old
* Has confirmed SARS-CoV-2 infection by RT-PCR method using sample collected from nasopharyngeal swab (NP) and oropharyngeal swab (OP) with Ct value in either one of the following cases

  1. Ct ≤ 26 if the subject has RT-PCR performed as part of screening procedures
  2. Ct ≤ 24 if the subject has had RT-PCR performed before admission and the time between the sample collection for RT-PCR and randomization is ≤ 24 hours
* Has been admitted for medical care at the investigational sites
* In case of symptomatic patient, date of symptoms onset is ≤ 7 days prior to randomization. In case of asymptomatic patient, the first date of positive result from RT-PCR or antigen test kit for SARS-CoV-2 is ≤ 7 days prior to randomization.
* Qualified for the criteria to receive favipiravir for COVID-19 treatment according to Guidelines on clinical practice, diagnosis, treatment, and prevention of healthcare-associated infection for COVID-19 in Thailand in either one of the following cases

  1. Will start receiving favipiravir during the study period or
  2. Has received favipiravir no more than 24 hours before receiving the investigational drug
* Asymptomatic or has mild to moderate COVID-19 as defined in section 7.2.2.
* Willing to participate in the study and able to provide written informed consent
* Women of childbearing potential must agree to either abstinence or use at least one primary form of contraception from the time of screening through D28.

Exclusion Criteria:

* Has severe or critical COVID-19 as defined in section 7.2.2.
* Bedridden (totally confined to bed)
* Has elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) over 3 times the upper range of normal limits, or history of liver cirrhosis
* Females only: Currently pregnant, as determined by positive β-human choriogonadotropin (HCG) test in urine, or breast-feeding
* Receiving other potential drugs for COVID-19 treatment prior to randomization including Remdesivir, Nitazoxanide, Chloroquine, Hydroxychloroquine, Azithromycin, Lopinavir-ritonavir, Famotidine, Tocilizumab, Baricitinib (except favipiravir)
* Received ivermectin within 1 month prior to the randomization
* Receiving other immunosuppressive or immunomodulatory drugs for the treatment of other conditions (not including topical steroids)
* History of hypersensitivity to ivermectin or favipiravir or any components of the drugs
* Receiving medications that increase gamma-aminobutyric acid (GABA) potentiating activity such as barbiturates, benzodiazepines, sodium oxybate, valproic acid, or receiving medications that prevent or inhibit the p-glycoprotein transport system such as amiodarone, carvedilol, clarithromycin, cyclosporine, erythromycin, itraconazole, ketoconazole, quinidine, ritonavir, tamoxifen, verapamil, amprenavir, clotrimazole, phenothiazines, rifampin, St. John's Wort etc.
* Has history of hereditary xanthinuria
* Has hypouricemia (serum uric acid ≤ 1 mg/dL), uncontrolled gout or history of xanthine urolithiasis
* Participating in other clinical trials or participated in other clinical trials in a period of one month or less than 5 half-lives of the study drug before screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
The rate of SARS-CoV-2 viral clearance | Day 1- Day 6
  The rate of viral clearance as measured by Ct values from NP and OP swab once daily

SECONDARY OUTCOMES:
Mortality rate | Day 14 and Day 28
  The proportion of subjects who died
Progression to severe disease | Day 1 to discharge Day, Day 14, Day 28
  The proportion of subjects with clinical deterioration by at least 2 points according to WHO ordinal scale for clinical improvement.
Duration of admission | Day 1 to discharge Day
  Number of days of admission
Oxygen requirement | Day 1 to Day 28
  * The proportion of subjects who require the use of supplemental oxygen, non-invasive oxygen supplementation, mechanical ventilation, extracorporeal membrane oxygenation (ECMO) and admission to the intensive care unit (ICU)
  * The duration that the subjects require the use of supplemental oxygen
Proportions of SARS-CoV-2 viral clearance | Day 6
  The proportion of subjects with negative RT-PCR for SARS-CoV-2

OTHER OUTCOMES:
Safety of ivermectin in combination with favipiravir | Day 1 to Day 28
  * The proportion of subjects who develop adverse events and serious adverse events associated with ivermectin.
  * The proportion of subjects who require discontinuation of ivermectin due to adverse events.
The effect of variants and viral genetic repertoires on investigational drug efficacy | Day 1
  Determination of correlation between genetic variants of SARS-CoV-2 and clinical manifestation/treatment efficacy among subjects
The inflammatory cytokine response | Day 1, 3, 5, discharge, and 28
  The reduction of plasma inflammatory cytokine levels during treatment
The immune response | Day 1 to Day 28
  The change of level of antibody and T cell response during treatment and follow up

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - JC Kevin Sathorn Bangkok Hotel, Bangkok
  - Songklanagarind Hospital, Bangkok